CLINICAL TRIAL: NCT02434016
Title: Assessing Diaphragm Muscle Inactivity in Mechanically Ventilated ICU Patients
Acronym: DIVIP
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB #15-073
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Insufficiency
Keywords: Diaphragm; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background: Mechanical ventilation is a life saving intervention in patients with acute respiratory failure, for instance, due to infection or trauma. The main goals of mechanical ventilation are to improve oxygenation and decrease the load imposed on the respiratory muscles. Unfortunately, mechanical ventilation comes with adverse events including disuse atrophy and weakness of the respiratory muscles. The diaphragm is the main muscle for inspiration and therefore this clinical entity is commonly referred to as ventilator-induced diaphragm dysfunction (VIDD). Several studies have shown that inspiratory muscle weakness is associated with adverse outcomes, including prolonged duration of mechanical ventilation. Inactivity or disuse is a recognized risk factor for the development of VIDD: disuse may result from excessive unloading of the diaphragm by the ventilator. Therefore, clinicians aim to limit the risk of VIDD by using ventilator modes that allow patients to perform at least part of the total work of breathing when deemed clinically appropriate. However, even when these so-called assisted modes for ventilation are used, excessive unloading of the diaphragm may occur; without using technology that allows monitoring of diaphragm function, the clinician is often uncertain as to whether this muscle is indeed actively working. Continuous recording of the electrical activity of the diaphragm (EAdi) is used to monitor diaphragm muscle activity in ICU patients. Furthermore, sonographic measurements of diaphragm thickness allows for an easy quantification of diaphragmatic activity (thickening fraction) as well as providing a potentially useful mechanism for studying diaphragm injury and function during mechanical ventilation.

Aim: To assess the duration of diaphragm muscle inactivity in patients admitted to the ICU using EAdi monitoring and to assess the correlation between diaphragm thicknening fraction, as measured by ultrasound, and electrical activity, as measured by EAdi.

Hypothesis: Diaphragm muscle inactivity frequently occurs in the early phase of ICU admission Design: Observational pilot study in ventilated adult ICU patients admitted to the ICU at St Michael's Hospital. The investigators aim to enroll 75 patients.

Primary outcome: Time from catheter positioning to first EAdi (> 5 uV last at least 5 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the ICU
* Intubation in the ICU or < 12 hours before admission
* Expected duration of mechanical ventilation > 48 h
* Edi monitoring tube / catheter in situ by the clinical team

Non-inclusion Criteria:

* Anticipated removal of EAdi tube within 48 hours of ICU admission (e.g., for MRI, for endoscopic intervention)
* High risk for intracranial hypertension or proven intracranial hypertension due to severe neurotrauma or substantial intracranial hemorrhage because these patients will likely need Magnetic Resonance Imaging. This can be discussed on a case-by-case basis based on the severity and initial findings
* Lack of Servo-i NAVA capable ventilator, lack of EAdi catheter

Exclusion Criteria:

* Phrenic nerve lesions (past medical history)
* Contraindications to the insertion of a naso- or oro-gastric (feeding) tube
* Patients already intubated for > 12 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the ICU in whom the attending clinician has decided to insert the dedicated feeding tube (EAdi catheter) in the ICU or < 12 hours before admission
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time from catheter positioning to first EAdi signal | Up to 5 days
  > 5uV lasting at least 5 minutes

SECONDARY OUTCOMES:
Time from endotracheal intubation to first EAdi signal | Up to 5 days
Time from catheter positioning until 24 hours of continuous EAdi signal | Up to 5 days
Number of patients without EAdi signal in the first 72 hours after intubation | Up to 3 days
Patient-ventilator interaction assessed by EAdi | Up to 5 days
Clinical characteristics associated with diaphragm inactivity | Up to 5 days
Correlation between diaphragm muscle thickness and diaphragm thickening fraction | Up to 5 days

OTHER OUTCOMES:
Correlation between the electrical activity of the diaphragm and diaphragm and intercostal thickening fraction | Up to 5 days
Correlation between thickening fraction of the intercostal muscles and of the diaphragm | Up to 5 days
Changes in diaphragm and intercostal muscle thickness over time | Up to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Laurent J. Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Sassoon CS, Zhu E, Caiozzo VJ. Assist-control mechanical ventilation attenuates ventilator-induced diaphragmatic dysfunction. Am J Respir Crit Care Med. 2004 Sep 15;170(6):626-32. doi: 10.1164/rccm.200401-042OC. Epub 2004 Jun 16. PMID 15201132
- [Background] Doorduin J, van Hees HW, van der Hoeven JG, Heunks LM. Monitoring of the respiratory muscles in the critically ill. Am J Respir Crit Care Med. 2013 Jan 1;187(1):20-7. doi: 10.1164/rccm.201206-1117CP. Epub 2012 Oct 26. PMID 23103733
- [Background] Heunks LM, Doorduin J, van der Hoeven JG. Monitoring and preventing diaphragm injury. Curr Opin Crit Care. 2015 Feb;21(1):34-41. doi: 10.1097/MCC.0000000000000168. PMID 25546533
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Derived] Sklar MC, Madotto F, Jonkman A, Rauseo M, Soliman I, Damiani LF, Telias I, Dubo S, Chen L, Rittayamai N, Chen GQ, Goligher EC, Dres M, Coudroy R, Pham T, Artigas RM, Friedrich JO, Sinderby C, Heunks L, Brochard L. Duration of diaphragmatic inactivity after endotracheal intubation of critically ill patients. Crit Care. 2021 Jan 11;25(1):26. doi: 10.1186/s13054-020-03435-y. PMID 33430930